CLINICAL TRIAL: NCT04930393
Title: A Randomized Double-blinded Study to Evaluate the Efficacy of PECS II Block Versus Intercostobrachial Ring Block in Patients Undergoing Arthroscopic Rotator Cuff Repair With Open Biceps Tenodesis
Brief Title: Evaluating the Efficacy of PECS II Block Versus Axillary Ring Block in Rotator Cuff Repair Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Paul S. Lee, Assistant Professor of Clinical Anesthesiology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HS-20-00980
Record Dates: First submitted 2021-04-28; First posted 2021-06-18 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient and Provider won't be aware of what block will be administered until just before the nerve block is done
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS II Block (Active Comparator): This group will receive an interscalene block in addition to a pectoral nerve block under ultrasound guidance with local anesthetic injected in the plane between the pectoralis minor and serratus anterior muscles
  Interventions: Procedure: Nerve Block - either PECS II or axillary ring
- Axillary Ring Block (Active Comparator): This group will receive an interscalene block in addition to a ring block with local anesthetic injected subcutaneously along the axilla from anterior to posterior direction.
  Interventions: Procedure: Nerve Block - either PECS II or axillary ring

INTERVENTIONS:
Procedure: Nerve Block - either PECS II or axillary ring — In addition to an interscalene nerve block, one of these two interventions will be administered to assess pain control after a biceps tenodesis

SUMMARY:
Our current standard of care is to perform an interscalene peripheral nerve block for patients receiving rotator cuff repair surgery as it is an effective opioid-free alternative for post-operative pain control. However, many of these repairs require a supplemental incision for an open biceps tenodesis, which is not covered by the interscalene block. The intercostobrachial nerve covers this incision and is targeted by an axillary ring block or a single shot nerve block in the fascial plane between the pectoralis minor and serratus anterior muscles (otherwise termed as a PECS II block). This study will attempt to delineate if one is superior in postoperative analgesia and mitigating intraoperative stimulation by comparing an axillary ring block to a PECS II block. Patients receiving a rotator cuff repair with biceps tenodesis without histories of chronic opioid use and respiratory compromise will be eligible to be enrolled in the study. All patients will receive an interscalene block and group 1 will receive a supplemental axillary ring block and group 2 will instead receive a PECS II block. After surgery, the patients' pain score will be assessed upon PACU arrival, at 6 hours after block, and 2 weeks postoperatively. Their opioid requirements will also be assessed. Our primary outcome is pain score at 6 hours following the block.

ELIGIBILITY:
Inclusion Criteria:

* medically optimized patients who will undergo an elective surgery for an arthroscopic rotator cuff repair with open biceps tenodesis

Exclusion Criteria:

* women who are pregnant or breastfeeding, history of chronic opioid use, respiratory compromise, smokers, or allergy to local anesthetics or opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score at 6 hours following the block | 6 hours post-block

SECONDARY OUTCOMES:
Morphine milligram equivalents (MME) | Right after surgery and 2 weeks
  MMEs in recovery room after surgery and 2 weeks after surgery via phone call
Intraoperative Stimulation | 2 hours during surgery
  Whether patient displayed signs of pain (movement, elevated blood pressure or heart rate) under moderate sedation in the operating room

CONTACTS AND LOCATIONS:
Locations (1):
- Healthcare Center 3 - Keck Hospital of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho CH, Song KS, Min BW, Jung GH, Lee YK, Shin HK. Efficacy of interscalene block combined with multimodal pain control for postoperative analgesia after rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2015 Feb;23(2):542-7. doi: 10.1007/s00167-012-2272-3. Epub 2012 Oct 30. PMID 23108685
- [Background] Liu XN, Noh YM, Yang CJ, Kim JU, Chung MH, Noh KC. Effects of a Single-Dose Interscalene Block on Pain and Stress Biomarkers in Patients Undergoing Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial. Arthroscopy. 2017 May;33(5):918-926. doi: 10.1016/j.arthro.2016.09.018. Epub 2016 Dec 14. PMID 27988164
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533
- [Background] Siddeshwara A, Singariya G, Kamal M, Kumari K, Seervi S, Kumar R. Comparison of efficacy of ultrasound-guided pectoral nerve block versus thoracic paravertebral block using levobupivacaine and dexamethasone for postoperative analgesia after modified radical mastectomy: A randomized controlled trial. Saudi J Anaesth. 2019 Oct-Dec;13(4):325-331. doi: 10.4103/sja.SJA_25_19. PMID 31572077
- [Background] Versyck B, van Geffen GJ, Chin KJ. Analgesic efficacy of the Pecs II block: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):663-673. doi: 10.1111/anae.14607. PMID 30957884
- [Background] Reynolds JW, Henshaw DS, Jaffe JD, Dobson SW, Edwards CJ, Turner JD, Weller RS, Graves BR, Freehill MT. Analgesic Benefit of Pectoral Nerve Block II Blockade for Open Subpectoral Biceps Tenodesis: A Randomized, Prospective, Double-Blinded, Controlled Trial. Anesth Analg. 2019 Aug;129(2):536-542. doi: 10.1213/ANE.0000000000004233. PMID 31136331